CLINICAL TRIAL: NCT07292415
Title: Nerve Grafting Using MATRIderm® in Traumatic Digital Nerve Injuries: a Randomized, Single-center, Controlled Study
Acronym: MATRINERVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-PP-12
Record Dates: First submitted 2025-12-01; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: This Study is Testing the Use of MatriDerm

STUDY DESIGN:
Intervention Model Description: 35 patients will receive standard nerve stitching alone. 35 patients will receive nerve stitching plus MatriDerm® wrapping.
Who Masked: Participant, Investigator
Masking Description: Researchers will evaluate finger sensation one year after surgery using standard touch tests. The hypothesis is that nerve wrapping with MatriDerm® will lead to better sensory recovery than stitching alone. By participating, patients will help improve treatments for hand injuries and support research on nerve healing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Nerve suture alone" group (Sham Comparator)
  Interventions: Procedure: Standard peripheral nerve repair under regional anesthesia with magnification; epineural sutures placed, followed by 2-week immobilization if needed.
- "Nerve suturing and sleeving" group (Experimental)
  Interventions: Procedure: Peripheral nerve repair under regional anesthesia with epineural sutures; nerve wrapped along its length with 1 mm MatriDerm® collagen-elastin matrix before standard skin closure.

INTERVENTIONS:
Procedure: Standard peripheral nerve repair under regional anesthesia with magnification; epineural sutures placed, followed by 2-week immobilization if needed. — Peripheral nerve repair will be performed in the operating room under axillary regional anesthesia, with a pneumatic tourniquet at 250 mmHg. The nerve will be exposed using a surgical microscope or magnifying loupes. The two nerve stumps will be carefully dissected, and epineural sutures will be placed using simple 9/10 stitches. When tension is present on the repair, postoperative immobilization will be applied for 2 weeks to protect the suture. Postoperative care and follow-up will be standardized, including regular assessments of sensory recovery and hand function.
  Arms: "Nerve suture alone" group
Procedure: Peripheral nerve repair under regional anesthesia with epineural sutures; nerve wrapped along its length with 1 mm MatriDerm® collagen-elastin matrix before standard skin closure. — Peripheral nerve repair will be performed in the operating room under axillary regional anesthesia with a pneumatic tourniquet at 250 mmHg. The nerve will be exposed using a surgical microscope or magnifying loupes. The two nerve stumps will be carefully dissected, and epineural sutures will be placed using simple 9/10 stitches, as in standard care. In addition, for patients in the MatriDerm® arm, the sutured nerve will be wrapped along the entire dissected length with a 1 mm MatriDerm® collagen-elastin matrix. The nerve and matrix will then be irrigated with saline before standard skin closure. Postoperative immobilization will be applied for 2 weeks if tension is present on the repair.
  Arms: "Nerve suturing and sleeving" group

SUMMARY:
Hand and wrist injuries are very common, with nearly 2 million cases each year in France. Many injuries involve cuts that damage important structures such as nerves, tendons, blood vessels, bones, or joints. About 12.5% of hand wounds affect nerves, which can cause numbness, pain, or abnormal nerve growths called neuromas. Patients may also experience unusual sensations or intolerance to cold.

The usual treatment for a cut nerve is to carefully stitch it back together. Sometimes, additional techniques can be used to help the nerve heal better and reduce scarring. One technique, called nerve wrapping, involves surrounding the damaged nerve with a small protective tube to support its repair.

This study is testing the use of MatriDerm®, a collagen-elastin matrix originally used to help skin heal. MatriDerm® acts like a scaffold, supporting tissue repair and controlling scar formation. Its properties may also help nerves heal when placed around a stitched nerve.

This is an academic, monocentric, prospective, randomized, controlled study conducted in a double-blind manner (neither the patient nor the evaluator knows which treatment is given). The goal is to see if wrapping a stitched nerve with MatriDerm® improves finger sensation recovery compared with stitching alone. Seventy patients with traumatic nerve injuries of the fingers will be included: one group of patients will receive standard nerve stitching alone and another group will receive nerve stitching plus MatriDerm® wrapping.

Researchers will evaluate finger sensation one year after surgery using standard touch tests. The hypothesis is that nerve wrapping with MatriDerm® will lead to better sensory recovery than stitching alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 16 to 75
2. Patient with a palm or finger wound with sensory nerve damage (partial >50% or total)
3. Indication for repair by direct suture in the operating room
4. Possibility of attending a follow-up visit after 1 year
5. Patient affiliated with a social security system
6. Patient who has given their written consent after receiving written and oral information

Exclusion Criteria:

1. Pre-existing sensory disorders
2. History of nerve damage in the affected hand
3. Known hypersensitivity to bovine proteins
4. Active infection in the affected hand
5. Patient protected by law under guardianship or curatorship, or unable to participate in a clinical study MATRINERVE 24-PP-12 Version No. 1.0 dated July 22, 2025 Page 8 of 40 clinical trial under Article L. 1121-16 of the French Public Health Code
6. Pregnant or breastfeeding women of childbearing age

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving ≤6 mm in 2-point static discrimination test at fingertip pulp 12 months after traumatic digital nerve repair, comparing MatriDerm® nerve wrapping versus standard nerve suturing. | 12 months after surgery (give or take 1 month)
  The primary outcome is the recovery of tactile discrimination in the fingertip pulp 12 months after surgery. It is assessed using the static 2-point discrimination test. The proportion of patients achieving a discrimination distance of ≤6 mm will be compared between the experimental group (nerve suturing plus MatriDerm® wrapping) and the control group (nerve suturing alone). This measure reflects the functional sensory recovery of the repaired nerve and allows evaluation of the potential benefit of MatriDerm® as an adjunct to standard nerve repair.

SECONDARY OUTCOMES:
Incidence of neuroma formation at 12 months after digital nerve repair | 12 months after surgery (give or take 1 month)
  The proportion of patients developing neuromas within 12 months after surgery will be compared between the experimental group (nerve suturing plus MatriDerm® wrapping) and the control group (nerve suturing alone). This measure evaluates whether MatriDerm® reduces the risk of neuroma formation after nerve repair.
Incidence of chronic pain at 12 months after digital nerve repair | 12 months after surgery (give or take 1 month)
  The proportion of patients reporting chronic pain one year after surgery will be compared between the experimental group (nerve suturing plus MatriDerm® wrapping) and the control group (nerve suturing alone). This measure assesses whether MatriDerm® reduces the occurrence of long-term postoperative pain.
Incidence of cold intolerance at 12 months after digital nerve repair | 12 months after surgery (give or take 1 month)
  The proportion of patients experiencing cold intolerance one year after surgery will be compared between the experimental and control groups. This measure evaluates the effect of MatriDerm® nerve wrapping on reducing postoperative sensitivity to cold.
Patient satisfaction with scar quality at 12 months after surgery | 12 months after surgery (give or take 1 month)
  Patient-reported satisfaction regarding the appearance and quality of the surgical scar will be collected using a 5-point scale (very satisfied, satisfied, neutral, disappointed, dissatisfied). Results will be compared between patients in the experimental group (MatriDerm® wrapping) and the control group (suture alone).
Overall patient satisfaction at 12 months after surgery | 12 months after surgery (give or take 1 month)
  Overall satisfaction with the surgical outcome will be assessed using a 5-point scale (very satisfied, satisfied, neutral, disappointed, dissatisfied). Comparison will be made between the experimental group (MatriDerm® wrapping) and the control group (suture alone) to evaluate the impact of MatriDerm® on overall patient satisfaction.